CLINICAL TRIAL: NCT06114069
Title: Prosthetic Management of All on Four Versus All on Six to Rehabilitate Completely Edentulous Maxillary Ridge Opposed by Natural Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr ELsaeed, researcher, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M07100522
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-08

CONDITIONS: Prosthesis Survival
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: The patients were classified into 2 groups:
  1. Group I; 4 patients received 4-implant supported fixed prosthesis.
  2. Group II; 4 patients received 6-implant supported fixed prosthesis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- all on four group (Active Comparator): 4 patients received 4-implant supported fixed prosthesis
  Interventions: Procedure: implant supported maxillary fixed prosthesis
- all on six group (Active Comparator): 4 patients received 6-implant supported fixed prosthesis
  Interventions: Procedure: implant supported maxillary fixed prosthesis

INTERVENTIONS:
Procedure: implant supported maxillary fixed prosthesis — Maxillary fixed prosthesis according to all on four or all on six concept

SUMMARY:
the aim of the study to compare the anterior maxillary bone index changes for patient rehabilitated with implant supported fixed prosthesis opposed by natural teeth

ELIGIBILITY:
Inclusion Criteria:

* 1. All patient wearing a maxillary implant supported overdenture or implant supported fixed restoration and mandibular natural teeth or fixed restoration within natural dentition.

  2. All patients were unsatisfied by the maxillary restoration and presented clear preference for a better prosthesis.

  3. They were healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetics or osteoporosis. This was achieved through medical history and clinical examination by physician.

  4. At least one year passed after the last restoration. 5. At least 15 mm restorative space must be available (from the mucosa covering the crest of the residual ridge to proposed occlusal plane) to permit construction of all types of tested prosthesis (class I according to Ahuja and Cagna).195 This was detected by a tentative jaw relation.

Exclusion Criteria:

* 1. Patients had head and neck radiotherapy, patients with bleeding disorders or hepatic patients.

  2. Patients with metabolic disorders as diabetes mellitus, osteoporosis and hepatic disorders which might affect implant lifespan.

  3. Long term immunosuppress and corticosteroid drug therapy. 4. Patient with abnormal habits as clenching and bruxism. 5. Smoking patient. 6. Uncooperative patients. 7. Neuromuscular diseases. 8. Patient with problems in TMJ.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
anterior area index | six months
  outcome is being evaluated by radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Saeed, Al Mansurah, DK, Egypt